CLINICAL TRIAL: NCT05543343
Title: Evaluating the Efficacy and Safety of Staphylococcus and Neisseria Tablets in the Treatment of Acute Exacerbations of Chronic Obstructive Pulmonary Disease.
Brief Title: Staphylococcus and Neisseria Tablets in the Treatment of Acute Exacerbations of Chronic Obstructive Pulmonary Disease.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qu Yiqing (Other)
Collaborators: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Qu Yiqing, Professor, Qilu Hospital of Shandong University
Organization: Qilu Hospital of Shandong University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: quyiqing@sdu.edu.cn
Record Dates: First submitted 2022-09-14; First posted 2022-09-16 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: COPD; Acute exacerbation; Bacterial lysates
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ntaphylococcus albicans tablets (Experimental): Participants received High-dose Staphylococcus albicans tablets (0.3 mg/tablet, 8 tablets each time, 3 times a day, Qilu Pharmaceutical Co., Ltd., course of treatment 90 days) or Normal-doseStaphylococcus albicans tablets (0.3 mg/tablet, 4 tablets each time, 3 times a day, Qilu Pharmaceutical Co., Ltd., course of treatment 90 days)+ placebo (4 tablets each time, 3 times a day, Qilu Pharmaceutical Co., Ltd., course of treatment 90 days).
  Interventions: Drug: High dose or normal dose staphylococcus albicans
- Placebo (Placebo Comparator): Participants received placebo (8 tablets each time, 3 times a day, Shandong Qilu Pharmaceutical Co., Ltd., course of treatment 90 days).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: High dose or normal dose staphylococcus albicans — 8 staphylococcus albicans tablets(0.3 mg) 3 times daily or 4 staphylococcus albicans tablets(0.3 mg)+4 placebo tablets 3 times daily
  Arms: Ntaphylococcus albicans tablets
Drug: Placebo — 8 placebo tablets 3 times daily
  Arms: Placebo

SUMMARY:
It is planned to enroll 495 acute exacerbation of chronic obstructive pulmonary disease patients, and they will be randomly assigned to the high-dose test group, normal dose test group or control group at a ratio of 1:1:1, with 165 patients in each group. The course of treatment is 90 days, and the total follow-up time is one year. The purpose of the study is to evaluate the effectiveness and safety of different doses of bacterial lysates (Staphylococcus and Neisseria Tablets) in the treatment of acute exacerbation of chronic obstructive pulmonary disease.

ELIGIBILITY:
Inclusion Criteria:

1. Age 40~75 years old (including both ends), gender is not limited；
2. Clinically diagnosed as chronic obstructive pulmonary disease (have a lung function test in the past year, after inhaling 400ug of salbutamol for 15 to 30 minutes, FEV1/FVC<0.70);
3. The patient was in the acute exacerbation of chronic obstructive pulmonary disease at the time of enrollment (the patient's cough, sputum expectoration, and dyspnea exceeded any abnormal variation);
4. At least one exacerbation of chronic obstructive pulmonary disease in the past year; The patient (or his legal representative) must sign and date the informed consent form, indicating that he/she understands the purpose of the study and the procedures to be carried out, and is willing to participate in the study.

Exclusion Criteria:

1. The investigator judges that the patient has serious diseases that are not suitable for inclusion in this study, including but not limited to the following diseases:

   1. Complicated with respiratory diseases that may affect the efficacy and safety evaluation of the experimental drugs (such as clinically significant: asthma, pneumonia, active tuberculosis, lung cancer, bronchiectasis, sarcoidosis, pulmonary fibrosis, pulmonary hypertension, interstitial lung diseases, cystic fibrosis, bronchiolitis obliterans, etc.);
   2. Complicated with a history of severe cardiovascular disease (such as: coronary artery insufficiency), clinically significant arrhythmia (such as high-grade atrioventricular block, atrial flutter/atrial fibrillation, supraventricular/ventricular tachycardia, etc.), hypertension, heart failure that cannot be effectively controlled, myocardial infarction occurred in the first 6 months before enrollment, or the results of the electrocardiogram have been judged by the investigator to have medical problems that may affect the safety of the patient;
   3. Complicated with other serious diseases or mental disorders (such as: stroke, epilepsy, uncontrolled hyperthyroidism, malignant tumors, etc.);
   4. Performed lobectomy, or performed lung volume reduction surgery within 12 months before screening;
   5. With multiple drug allergies;
   6. Alcoholism or drug abuse;
   7. Participated in other clinical studies within 3 months;
   8. End-stage COPD patients;
   9. Previously (within 6 months before the start of the study) or currently taking immune stimulating drugs at the same time (including thymosin, interferon, transfer factor, BCG polysaccharide, pneumonia vaccine and any kind of bacterial extracts, such as Biostim, except influenza vaccine) or immunization inhibitor
2. During the acute exacerbation hospitalization, use intravenous hormone for more than 7 days and/or continuous hospitalization for more than 15 days;
3. Have fertility and have not taken effective contraceptive measures (contraceptive methods include barrier contraception or hormonal contraception; barrier contraception includes: cervical cap, condom, intrauterine device, vaginal sponge, spermicide; hormonal contraception includes: contraceptive) ； According to the judgment of the investigator, the patient is not suitable for research observation.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 495 (Estimated)
Dates: Start 2022-01-05 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Number of acute exacerbations of chronic obstructive pulmonary disease in 1 year | From enrollment to the end of the 1-year follow-up period
  The number of acute exacerbations of COPD in one year since the patients were enrolled in the group.

CONTACTS AND LOCATIONS:
Overall Officials: Yiqing Qu, Study Chair — Qilu Hospital of Shandong University
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No